CLINICAL TRIAL: NCT00632112
Title: A Real Life Evaluation of the Performance of a Large Volume Nebulizer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Arkansas Children's Hospital Research Institute (Other)
Collaborators: S&T Medical Technologies, Inc. (Industry)
Responsible Party: Ariel Berlinski, University of Arkansas for Medical Sciences
Other Study IDs: 98551
Record Dates: First submitted 2008-02-29; First posted 2008-03-10 (Estimated); Last update posted 2009-06-05 (Estimated); Status verified 2009-06

CONDITIONS: Asthma
Keywords: large volume nebulizer
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Continuous albuterol has become the standard of care for patients in status asthmaticus. We have previously performed an in-vitro study comparing 4 different brands of continuous nebulizers. We now want to compare the in-vitro with the in-vivo performance of the brand we use. we hypothesize that there will be no difference between in-vivo and in-vitro results.

DETAILED DESCRIPTION:
There will be no intervention to the patients. Nebulizers will be used as per current policies and procedures. They will only be marked on the outside at the water level every 2 hours for the first 6 hours. Once ready to be discarded will be collected for laboratory testing Once in the laboratory, nebulizers will be weight on a precision scale without liquid, then they will be filled with normal saline to the first mark (6th hour) and re-weight. The nebulizers will be filled to next mark and re-weight until 200 mls. of total volume are achieved. Solution output will be calculated as the weight difference between the 2 hour periods.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients admitted to Pediatric Intensive Care Unit due to status asthmaticus, requiring continuous albuterol nebulization.

Exclusion Criteria:

* Patients requiring invasive or non-invasive ventilation.

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric patients admitted to the Pediatric Intensive Care Unit due to status asthmaticus, requiring continuous albuterol nebulization.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2008-03; Primary Completion 2009-07 (Estimated)

PRIMARY OUTCOMES:
Nebulizer solution output | every 2 hours for first 6 hours

CONTACTS AND LOCATIONS:
Overall Officials: Ariel Berlinski, M.D., Principal Investigator — University of Arkansas
Locations (1):
- Arkansas Children's Hospital, Little Rock, Arkansas, United States